CLINICAL TRIAL: NCT05453227
Title: Zinc Containing Vaginal Topical " Suppository " in Improving Post Menopausal Genitourinary Syndrome: "Double Blind Controlled Study "
Brief Title: Zinc Containing Vaginal Topical " Suppository "
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Bahaa Mohamed
Record Dates: First submitted 2022-06-21; First posted 2022-07-12 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Genitourinary Syndrome of Menopause
MeSH Terms: interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc Group (Active Comparator): 25 cases will be undergo treatment with active ingredient
  Interventions: Drug: Zinc
- Plcebo Group (Placebo Comparator): 25 cases will be undergo treatment with placebo
  Interventions: Drug: Zinc

INTERVENTIONS:
Drug: Zinc — To test the effect of a novel zinc-containing vaginal topical on GSM/VVA symptoms.

SUMMARY:
The genitourinary syndrome of menopause (GSM) is a new term that describes various menopausal symptoms and signs associated with physical changes of the vulva, vagina, and lower urinary tract.

The GSM includes not only genital symptoms (dryness, burning, and irritation) and sexual symptoms (lack of lubrication, discomfort or pain, and impaired function), but also urinary symptoms (urgency, dysuria, and recurrent urinary tract infections [UTI])

DETAILED DESCRIPTION:
The terms vulvovaginal atrophy and atrophic vaginitis were widely used until recently, but they have been considered to be inadequate for referring to the constellation of symptoms and signs associated with the genitourinary system after menopause.

The term vulvovaginal atrophy mentions the vulva and vagina only, and these words are not used comfortably in general social discussion and in the media. The term atrophic vaginitis implies a state of inflammation or infection, which is not a primary component of menopausal changes. In addition, a limitation of the terms vulvovaginal atrophy and atrophic vaginitis is that they do not take into account the symptoms of the lower urinary tract, which are among the most important symptoms related to menopause.

Vulvovaginal atrophy (VVA) is a prevalent condition affecting many postmenopausal women.1 Up to 40% of postmenopausal women develop symptoms of VVA.

It is most often diagnosed by its symptoms, including vaginal dryness, burning, itching, vagina pain and dyspareunia. More recently these symptoms have been described as a syndrome: the genitourinary syndrome of menopause (GSM).

This new term describes various menopausal symptoms and signs including not only genital symptoms but sexual (pain) and urinary symptoms (dysuria, urgency) as well.

The pathophysiology of GSM/VVA can be explained by the decline in estrogen levels associated with diminished ovarian function and natural aging.

Traditionally the treatment options for GSM/VVA was vaginal estrogen supplementation but many women are either unable to or are afraid to use hormones. There are several non-hormonal treatment modalities for the management of VVA related symptoms, especially for one of the most bothersome symptoms of vaginal dryness.

The 2013 position statement of The North American Menopause Society indicates that the first-line therapies to alleviate symptoms of VVA should include non-hormonal vaginal lubricants and moisturizers as well as regular sexual activity.

Although there are numerous vaginal moisturizers and lubricants are commercially available only a few of those have been tested in clinical trials.

Previously the investigators showed the role of vaginal zinc supplementation on vaginal remodeling. The investigators showed that in human vaginal smooth muscle cells, zinc has a beneficial effect on the production of extracellular components produced by the muscle at 20 μM zinc tissue level, thereby increasing the amount of elastin production.

Earlier animal studies have shown that zinc plays an important role in the vaginal extracellular matrix (ECM) composition. When rats were kept on a zinc-lacking diet, the vaginal structure became similar to the menopausal vagina.With vaginal zinc replacement, the vaginal ECM could be regenerated with characteristics equivalent to juvenile rats .

ELIGIBILITY:
Inclusion Criteria:

* presence of symptoms of vulvovaginal atrophy/GSM in postmenopausal women. including vaginal dryness, burning, itching, vagina pain and dyspareunia. To be defined as a postmenopausal woman.

individuals had to have at least 12 consecutive months of amenorrhea without any other obvious reason/or consistently elevated follicle-stimulating hormone blood levels of 30 mIU/mL or higher.

Exclusion Criteria:

* premenopausal state,
* local or systemic hormone therapy within the past six months
* vaginal infection at presentation
* cytological atypia
* prior radiation treatment
* history of breast, ovarian or other gynecological cancer
* pelvic organ prolapse > stage 2
* recent use (3 months) of any vaginal product or douching.

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The using of novel zinc-containing vaginal suppositories | From baseline to 2 weeks after using the zinc sulphate
  Assessment of postmenopausal symptoms as dryness, burning, and irritation by Vaginal Health Index (VHI) score: elasticity, fluid secretion, pH and epithelial mucosa (integrity) and moisture components. Each component is scored on a scale of 1 (worst) to 5 (best). Lower scores indicate more severe atrophy. VHI was calculated at baseline and 2 weeks after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Assem Anwar, Professor, Study Chair — Department of Obstetrics & Gynecology Faculty of Medicine for boys, Al-Azhar University
Locations (1):
- Al-Azhar University Hospitals and Ashmoun central hospital, Cairo, Elmenofia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided